CLINICAL TRIAL: NCT02903264
Title: Gestational Diabetes Mellitus, Obesity and Periodontal Disease: a Cross Sectional Study
Brief Title: Gestational Diabetes Mellitus, Obesity and Periodontal Disease
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carla Andreotti Damante, Associate professor, University of Sao Paulo
Other Study IDs: BauruSchoolDentistry
Record Dates: First submitted 2016-09-06; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus, Gestational; Periodontal Diseases; Obesity
Keywords: Gestational Diabetes Mellitus; Obesity; Periodontal Disease
MeSH Terms: conditions — Diabetes, Gestational; Periodontal Diseases; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- GDM group: Gestational diabetes mellitus patients under treatment of an endocrinologist
  Interventions: Other: Gestational diabetes mellitus
- Control: Healthy non-pregnant females

INTERVENTIONS:
Other: Gestational diabetes mellitus
  Groups: GDM group

SUMMARY:
This study evaluated the periodontal condition of gestational diabetes mellitus (GDM) patients and a healthy non-pregnant control group. For the GDM group all medical data were recorded, including obesity/insulin resistance indicators.

DETAILED DESCRIPTION:
Gestational diabetes mellitus is associated to a worse periodontal condition. Many patients with these two diseases are also obese. After delivery, some patients maintain the pre-pregnancy obesity status and this condition is also associated to periodontal disease. The mechanisms involved in the relationship of all these medical and periodontal conditions are not clear.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for GDM group was pregnant women with diagnosis of GDM based on glucose determination described in a previous study (19) and under medical treatment of an endocrinologist and the presence of at least one tooth per sextant.
* Inclusion criteria for control group were absence of periodontal disease, mean age similar to test group and presence of at least one tooth per sextant.

Exclusion Criteria:

* The exclusion criteria for GDM group were pregnant women without diagnosis of diabetes, age below 18 years or higher than 42 years, and the presence of other systemic diseases.
* In control group, women were excluded if they were pregnant, had diabetes or other systemic disease and age below 18 years or higher than 42 years.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Only female participants
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2007-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Periodontal disease (gingivitis and periodontitis) measured by a periodontal probe and classified according to severity | One day
  Severe periodontitis was defined by the presence of ≥ 2 interproximal sites in different teeth with CAL ≥ 6mm and ≥1 interproximal site with PPD ≥5mm. Moderate periodontitis was defined by the presence of ≥ 2 interproximal sites in different teeth with CAL ≥ 4mm or ≥ 2 interproximal sites in different teeth with PPD ≥5mm. Mild periodontitis was defined as ≥ 2 interproximal sites in different teeth with ≥ 3 mm CAL and ≥ 2 interproximal sites in different teeth with ≥ 4 mm PPD or at least 1 site with PPD ≥ 5 mm (20,21). Gingivitis was determined as follows: Subjects were considered healthy if presented PPD ≤3mm/BOP extent scores < 10% and with gingivitis if presented PPD ≤3mm/ BOP extent scores >10%. Prevalence of periodontal disease was the sum of gingivitis, mild, moderate and severe periodontitis.
Obesity measured by a tape and a scale | one day
  Obese if: body mass index - BMI ≥ 25 Kg/m2 (weight in kilograms, height in meters) Obese if : waist-to-hip ratio - WHR >0.85 (cm)
Gestational diabetes mellitus diagnosed by an endocrinologist | one day
  Diagnosis stablished by a doctor based on glucose determination. The data was registered in the patient's medical chart.

SECONDARY OUTCOMES:
Dyslipidemia as an indicator of obesity/insulin resistance | one day
  The data was registered in the patient's medical chart. Dyslipidemia = HDL ≤ 35 mg/dL / LDL≥ 100 mg/dL / Total cholesterol ≥200 mg/dL / Triglycerides ≥ 150 mg/dL / VLDL < 30 mg/dL
Leukocytosis as an indicator of inflammation | one day
  The data was registered in the patient's medical chart.
  ≥ 10.000/L

CONTACTS AND LOCATIONS:
Overall Officials: Carla Damante, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Bauru School of Dentistry, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xie Y, Xiong X, Elkind-Hirsch KE, Pridjian G, Maney P, Delarosa RL, Buekens P. Prepregnancy obesity and periodontitis among pregnant females with and without gestational diabetes mellitus. J Periodontol. 2014 Jul;85(7):890-8. doi: 10.1902/jop.2013.130502. Epub 2013 Dec 19. PMID 24354652